CLINICAL TRIAL: NCT01093742
Title: A Dose Block-randomized, Double-blind, Placebo-controlled, Single Dosing, Dose-escalation Phase I Clinical Trial to Investigate the Safety, Tolerability and Pharmacokinetics of HM10560A After S.C. Administration in Healthy Male Subjects
Brief Title: A Study of HM10560A in Healthy Male Subject
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: HM-GHA-101
Record Dates: First submitted 2010-03-25; First posted 2010-03-26 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2014-02

CONDITIONS: Healthy
Keywords: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- cohort 1 (Experimental): HM10560A 0.089 mg/kg or Placebo
  Interventions: Drug: HM10560A; Drug: Placebo
- cohort 2 (Experimental): HM10560A 0.179 mg/kg or Placebo
  Interventions: Drug: HM10560A; Drug: Placebo
- cohort 3 (Experimental): HM10560A 0.357 mg/kg or Placebo
  Interventions: Drug: HM10560A; Drug: Placebo
- cohort 4 (Experimental): HM10560A 0.714 mg/kg or Placebo
  Interventions: Drug: HM10560A; Drug: Placebo

INTERVENTIONS:
Drug: HM10560A — Subcutaneously administrate at 0 hour on Day 1
Drug: Placebo — Placebo

SUMMARY:
* Study Design

  * Randomized, Double-blind, Placebo-controlled, escalating single-dose design.
  * Four ascending dose cohorts.
  * In each cohort, subjects will be randomized to receive a single dose of HM10560A or placebo (negative control).
* Objectives

  * The primary objective of the study is to assess the safety and tolerability of single escalating subcutaneous doses of HM10560A in healthy male subjects.

DETAILED DESCRIPTION:
The secondary objectives of the study are as follows:

* To assess the pharmacokinetics(PK) and pharmacodynamics(PD) of a single subcutaneous dose of HM10560A.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male volunteers, age range 20 to 54 years are informed of the investigational nature of this study and voluntarily agrees to participate in this study
2. Body mass index of ≥19 and ≤26 Subject
3. Medically healthy with no clinically significant screening results through Physical examination, 12 lead ECG, Laboratory test
4. Able to participate in all procedure
5. SBP 90-140 mmHg, DBP 60-90 mmHg, Pulse rate 50-90 times/min
6. AST, ALT <1.5 X UNL, CPK < 2 X UNL
7. Able to abstain from alcohol and smoke during study period
8. Consented to contraception until 2 month after end of the study

Exclusion Criteria:

1. Acute infection history within 14 days
2. Prior exposure or hypersensitivity to recombinant human growth hormone
3. Positive findings on HBsAg, Anti-HAV IgM, anti-HCV, HIV Ag, HIV Ab and syphilis high quality regain test
4. History of significant gastrointestinal, cardiac, pulmonary, hepato- and nephro- disease
5. psychiatric disorder, malignancy tumor, hormonal disorder, diabetes mellitus and hypertension or history of immunosuppressant treatment
6. Caffeine, alcohol and smoke abuse
7. History of hemophilia or anticoagulant treatment
8. Revulsion and/or panic about syringe needle and hypersensitivity to subcutaneously administration
9. History drug abuse or positive testing for amphetamine, barbiturate, cocaine, opiates, benzodiazepines
10. Blood donation or significant blood loss within 60 days prior to Day 1. Plasma donation or transfusion within 30 days prior to Day 1.
11. Receipt of another investigational medication within 60 days prior to Day 1
12. Use of any herbal products within 30 days or prescription medication within 14 days or over-the-counter medication within 7 days prior to the Day 1.
13. Subjects who are unlikely to comply with the protocol requirements, instructions and study related restrictions

Ages: 20 Years to 54 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2010-03; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Safety | 1, 2, 3, 5, 7, 11, 15, 22, 29 day after administration
  Investigate Safety of HM10560A:
  * Physical examination, Laboratory test, ECG, Vital sign, Adverse event, Local tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Jahon Kang, Study Director — Hanmi pharma.
Locations (1):
- Medical Center, Seoul, South Korea